CLINICAL TRIAL: NCT03165448
Title: Validation of Universal Scale in Oral Surgery (USOS) for Patient's Psycho-emotional Status Rating
Status: Completed | Type: Observational
Sponsor: Inesa Astramskaitė (Other)
Responsible Party: Sponsor-Investigator, Inesa Astramskaitė, Principal investigator, Lithuanian University of Health Sciences
Organization: Lithuanian University of Health Sciences (Other)
Other Study IDs: USOS validation
Record Dates: First submitted 2017-05-21; First posted 2017-05-24 (Actual); Last update posted 2017-05-24 (Actual); Status verified 2017-05

CONDITIONS: Fear, Dental
Keywords: oral surgery; psychology; fear; pain; dentistry
MeSH Terms: conditions — Pain

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Self-reported questions: All the participants will enroll the same study protocol, without any exceptions: pre-operative patient's self-reported questioning, post-operative doctor's questioning, 4-6 weeks patients retesting.
  Interventions: Diagnostic Test: Pre-operative USOS scale testing; Diagnostic Test: Pre-operative SDPQ, MDAS and VAS testing; Diagnostic Test: Post-operative doctor's reported USOS; Diagnostic Test: Re-testing 4-6 weeks later

INTERVENTIONS:
Diagnostic Test: Pre-operative USOS scale testing — Patient has to self-report USOS questionnaire just before the procedure as main scale.
Diagnostic Test: Pre-operative SDPQ, MDAS and VAS testing — Patient has to sel-report SDPQ, MDAS and VAS questions as control scales.
Diagnostic Test: Post-operative doctor's reported USOS — Operating doctor has to fill the USOS doctor's part o questionnaire just after the procedure.
Diagnostic Test: Re-testing 4-6 weeks later — All the participants has to refill USOS questionnaire 4-6 weeks later.

SUMMARY:
Patient's psycho-emotional status is being affected during various dental procedures causing patient's and doctor's discomfort. There are three basic factors, composing psycho-emotional status: fear, stress and pain sensitivity. There aren't any objective method that may help in standard evaluation of oral surgery patient's psycho-emotional status. In the present non-standardized evaluation, there is a problem of heterogeneity between studies, and also ineffective patient's evaluation. Therefore, Universal Scale in oral surgery for patient's psycho-emotional status rating (USOS) was designed. Clinical trial to validate the USOS was constructed.

DETAILED DESCRIPTION:
Patient's discomfort ant doctor's negative emotional feelings in various dental procedures are related to patient's psycho-emotional status during the procedure. Three main factors, determining patient's psycho-emotional status, were determined in earlier studies: fear, stress and pain sensitivity.

Different elements cause patient's fear, stress and pain sensitivity, therefore in order to improve patient's psycho-emotional status, the causative element should be known. Multifactority o human's psycho-emotional status is described by anatomy - emotional state depends on amygdala (lat. corpus amygdaloideum) and cerebellum (lat. cerebellum), which interaction is related to development of fear to negative irritants. This process arise from two steps learning system - negative experience may cause fear and corresponding reactions. Dejean et al stated, that the main locations, in which memories causing fear are kept, are in dorsomedial prefrontal cortex. In this area 4Hz frequency vibrations are found during the fearful reactions. Neurologic examinations prove that emotional-physical relationships are firm and negative emotions may cause various reactions in organism. However, changes caused by fear, that are found in brain, are not specific. Various emotions may cause different vibrations in specific recurrent cortex locations, therefore it is important to rate full psycho-emotional status complex.

When the present of fears and phobias were examined, fear to dental treatment is in top-5 of all fears and in phobias - it is number one. The strength of dental fear may vary according to the upcoming procedure. Oosterink et al found that out of 67 dental procedures, oral surgery is the most terrifying for patients. When only oral surgery procedures were examined, third molar extraction was found as most fear producing.

Pain sensitivity - the other important part of patient's psycho-emotional status, which is described as patient's painful reaction to minimal stimulus and opportunity to maintain the maximum pain. Even though the pain is usually described as reaction to physical stimulus, it is closely related to patient's psychology. Previous pain experience may generate negative memories, which cause more sensitivity in repeated procedure. Also, it is known that stronger pain may be felt if it was expected before. Only physical methods to control the pain are not always effective - patient's psycho-emotional status correction is needed in better control of pain, which can be achieved with non-interventional methods.

Stress is usually described as physical reactions provoked by negative stimulus, which arise with active sympathetic nervous system and behavioral changes. It should be noted, that fear and felt pain may cause stress. Also, it was found that long term felt stress may cause chronic pains evaluations and vice versa - any pain felt provokes stressful reactions in human's body. Therefore, stress as physiological reactions arise because of painful interventions, same as for physiological fear - stimuli, that are constantly present during oral surgery procedures.

Nowadays there are various medication and non-medication methods to control patient's fear, stress and pain sensitivity in dental procedures. However, in order to examine effectivity of these methods and overall the problem of patient's psycho-emotional status, measures are needed. In earlier studies it was found that various general instruments are used to rate patient's fear and anxiety before teeth extraction procedures. Because of non-standardized rating, studies because such heterogeneous, that the results are incomparable between each other. The use of different questionnaires often showed different results even in the same situations. Because of their properties and actuality of the problem, there is a need to standardize patient's psycho-emotional status evaluation methods, with a use of practically adaptable measures.

Universal Scale in Oral Surgery (USOS) for patient's psycho-emotional status evaluation, composed from patient's reported part and doctor's reported part, was designed in earlier study by authors. The aim of present study is to assess the clinical effectivity and validate the USOS in case of outpatient tooth extraction for adult healthy patients.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients (18 years and more), who need routine tooth extraction
* No contraindications for outpatient tooth extraction
* Tooth extraction with local anesthesia
* Voluntary participation in the study
* Patients, that can fill questionnaires and enroll in the study by selves

Exclusion Criteria:

* Under-age patients and adult patients, who need inpatient tooth extraction
* Contraindications for outpatients tooth extraction
* Tooth extraction with general anesthesia or sedation
* Disagreement of participation in study
* Patients, that were unable to fill questionnaires and enroll the study by selves

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Healthy adult patients that came to Lithuanian university o health sciences, Department o oral and maxillofacial surgery clinic or outpatient tooth extraction were randomly selected.
Sampling Method: Probability Sample
Enrollment: 90 (Actual)
Dates: Start 2016-05-01 (Actual); Primary Completion 2016-12-01 (Actual); Study Completion 2017-04-01 (Actual)

PRIMARY OUTCOMES:
Correlation between USOS and control scales | The same day of the tooth extraction procedure
  The correlation degrees between USOS mean values and control scales mean values will be calculated.
Correlation between patient's and doctor's results | The same day of the tooth extraction procedure
  Correlations between patient's USOS part and doctor's USOS part will be calculated.
Re-testing o USOS | At 4-6 weeks time period, when USOS is being re-tested
  Correlation between USOS and re-tested USOS 4-6 weeks later will be calculated.

SECONDARY OUTCOMES:
Sex influence on patient's psycho-emotional status | The same day of the tooth extraction procedure
  The differences among men and women will be observed
Age influence on patient's psycho-emotional status | The same day of the tooth extraction procedure
  The differences between people with different age will be observed
Experience influence on patient's psycho-emotional status | The same day of the tooth extraction procedure
  Calculations, weather injectional anesthesia and oral surgery procedures experience influence the outcomes, will be performed

IPD SHARING:
Plan to Share IPD: No
Individual participants data is not important or study outcomes and will not be shared in any circumstances.